CLINICAL TRIAL: NCT05685082
Title: Teaching the Social Determinants of Health to Nursing Students With Culturally Diverse Simulation: A Quasi Experimental Trial
Brief Title: Teaching the Social Determinants of Health to Nursing Students With Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Semiha Asli Bozkurt, Principal investigator, University of Massachusetts, Boston
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BOZKURT-Int-001
Record Dates: First submitted 2022-12-22; First posted 2023-01-13 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Simulation of Physical Illness; Nurse's Role
Keywords: Nursing student; Simulation-based training; Standardized patient simulation; Manikin-based simulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized patient group (Experimental): The standardized patient simulation participants will receive a simulation with standardized patients on how to identify social determinants of health in an individual
  Interventions: Behavioral: Standardized patient simulation
- Manikin-based group (Experimental): The manikin-based simulation participants will receive a simulation with manikins on how to identify social determinants of health in an individual
  Interventions: Behavioral: Manikin-based simulation

INTERVENTIONS:
Behavioral: Standardized patient simulation — The standardized patient simulation participants will receive a simulation with standardized patients on how to identify social determinants of health in an individual
  Arms: Standardized patient group
Behavioral: Manikin-based simulation — The manikin-based simulation participants will receive a simulation with manikins on how to identify social determinants of health in an individual
  Arms: Manikin-based group

SUMMARY:
The goal of this intervention study is to compare two different simulation modalities (standardized patient and manikin-based) in nursing student education. The main aim is to determine the effect of new scenarios on cultural awareness levels in two different types of simulation modalities and to determine the effect of new scenarios on social determinants of health knowledge levels in two different types of simulation modalities.

Participants will assign to two groups and will attend simulation sessions.

DETAILED DESCRIPTION:
The simulation session will contain prebriefing, simulation, and debriefing. The participants will be assigned to the simulation session.

* The first group will be the standardized patient group. They will ask to fill out the Cultural Awareness Scale and social determinants of health knowledge. Then, they will attend prebriefing, standardized patient simulation, and debriefing.
* The second group will be the manikin-based group. They will ask to fill out the Cultural Awareness Scale and social determinants of health knowledge. Then, they will attend prebriefing, manikin-based simulation, and debriefing.

ELIGIBILITY:
Inclusion Criteria:

* being enrolled in Nursing in the Community course
* accepting to be a participant
* accepting to be recorded

Exclusion Criteria:

* not attending at least one of the prebriefing, simulation, or debriefing sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline cultural awareness level on the 36 questions Cultural Awareness Scale | Three hour
  The Cultural Awareness Scale is a validated, reliable, and self-reported instrument assessing cultural awareness levels. Each statement is graded from 1=Strongly Disagree to 7=Strongly Agree. While lower scores indicate less cultural awareness, higher scores indicate greater cultural awareness (minimum = 36, maximum = 252).
Change from baseline social determinants knowledge on the 10 questions Social Determinants of Health Survey | Three hour
  Social Determinants of Health Survey is a 10-question multiple-choice survey created by researchers by searching the literature. The number of responses to the answer choice is determined. The lower scores indicate fewer social determinants of health knowledge and higher scores indicate greater social determinants of health knowledge (minimum = 0, maximum = 10).

CONTACTS AND LOCATIONS:
Overall Officials: Semiha Asli Bozkurt, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No